CLINICAL TRIAL: NCT05834530
Title: Electromyographic Activity, Accuracy, Patient Satisfaction and Retention of Conventional Versus 3-D Printed Maxillary Complete Denture: A Cross-over Randomized Controlled Trial
Brief Title: Comparison of Conventional Versus 3-D Printed Complete Denture Regarding Retention, Accuracy, Elctromyographic Activity and Patient Satisfaction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Shereen Kabeel, Associate Professor, Al-Azhar University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: REC-PD-22-21
Record Dates: First submitted 2023-01-22; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Edentulous Mouth
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Complete Denture (No Intervention)
- 3 D printed Complete Denture (Experimental)
  Interventions: Other: 3D Printed Complete Dentures

INTERVENTIONS:
Other: 3D Printed Complete Dentures — Denture bases printed from a pre-polymerized block via additive technique, using photon S desktop 3D printer* that relies on SLA technology and post cured by post curing unit.
  Arms: 3 D printed Complete Denture

SUMMARY:
Analyzing and comparing the retention, accuracy, EMG and patient satisfaction of maxillary complete denture base fabricated by conventional and rapid prototyping techniques.

ELIGIBILITY:
Elligibility Criteria:

Inclusion Criteria:

* Completely edentulous patients were selected to have their ridges covered with firm, thick and compressible mucosa
* All patients accepting prosthodontic treatment by an removable denture.

Exclusion Criteria:

* TMJ disorder.
* Limited mouth opening or mandibular movement
* Muscle spasm or tenderness
* Mandibular deviation

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change of Retention | 3 months
  Retention was measured for both groups using the universal testing machine. Modification in each denture was made where two small metal tubes (3 mm diameters) were placed a few millimeters above the laterals in maxillary dentures by self-cure acrylic resin. The distance between the right tube and the geometric center was almost the same distance as between the left tube and the geometric center. The exact distance was checked using an orthodontic wire.

OTHER OUTCOMES:
Accuracy | up to 1 week
  The fitting surfaces of each upper denture was sprayed and scanned after finishing and before delivery, then was saved as an STL file after flipping of the denture's fitting surface to resemble the cast surface. Geomagic software was used to evaluate the accuracy at which the master cast STL file was selected as a reference data and the STL file of the flipped fitting surface of the denture was selected as a measured data. Both files were automatically aligned together by selecting the "best fit alignment "icon. The accuracy of the denture bases generated in a color map according to the 3D deviation between the denture base and reference data. Blue color indicates negative deviation (tissue compression), yellow to red color indicates positive deviation (misfit with space) while green color indicates measured deviation below 0.2mm.
Electromyography Change | 3 months
  The electromyographic activity was recorded for each patient by Nemus 2 machine. Washing period of 2 weeks between each denture as the same in masticatory efficiency and recorded as follow: The electromyographic activity was performed by measuring muscle activity of the masseter muscle on both sides
Change of Patient satisfaction | 3 months
  Patient satisfaction was investigated through a questionnaire, which was given to the patients. Evaluation of patient satisfaction was measured using the visual analogue scale (VAS) in which patients scored their answers using a scale from 0 to 10 cm (low/worst to high/best).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, AlAzhar University for Girls, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided